CLINICAL TRIAL: NCT04668924
Title: Prospective Evaluation of Photorefractive Intrastromal Crosslinking (PiXL) Without Epithelium Debridement (Epi-on) in High Oxygen for Progressive Keratoconus.
Brief Title: Epi-on PiXL for the Treatment of Progressive Keratoconus.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIXLKC-II
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Keratoconus; Corneal Crosslinking; Corneal Densitometry; Scheimpflug Photography; Corneal Disorder; Eye Diseases
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epi-on PiXL in high oxygen (Experimental): Photorefractive intrastromal corneal crosslinking without epithelium debridement during humidified high oxygen flow.
  Interventions: Procedure: Epi-on PiXL in high oxygen

INTERVENTIONS:
Procedure: Epi-on PiXL in high oxygen — After local anaesthetics, the keratoconus cornea is soaked in Riboflavin by repeated topical application during 10 minutes. A Riboflavin soaked sponge is used to lightly disrupt the epithelium tight junctions, without epithelium debridement. The cornea is illuminated with PiXL under 16:40 minutes during continuously delivery of humidified high oxygen via specific oxygen googles. The UV-dosage is individually customized based upon Kmax; for < 45 Diopters (D) 7.2J/cm^2 will be used; for 45-50D 10J/cm^2 will be used; for > 50D 15 J/cm^2 will be used.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and postoperative ocular discomfort by individually customized Photorefractive intrastromal crosslinking (PiXL) without epithelium debridement in high oxygen environment (Epi-on) for progressive Keratoconus.

DETAILED DESCRIPTION:
The study is designed as a prospective, open-label, nonrandomized trial involving participants of both genders aged 18-35 years with Keratoconus planned for routine corneal crosslinking at the Department of Ophthalmology, Umeå University Hospital, Umeå, Sweden.

The study includes 30 participants with unilateral Keratoconus, receiving Epi-on PiXL in high oxygen environment (n=30). All patients are informed about the procedures before consenting to participate in the study.

At baseline, before treatment, each eye is examined with slit-lamp microscopy, subjective refraction, determination of uncorrected (UCVA), low contrast visual acuity at 2.5 percentage contrast and 10 percentage contrast and best corrected (BSCVA) visual acuities using the LogMAR fast protocol and intraocular pressure (IOP) using Goldmann applanation tonometry. Under standardized, mesopic light conditions each eye is evaluated by keratometry readings and central corneal thickness, extracted from Schemipflug camera measurements, Pentacam HR® (Oculus, Inc. Lynnwood, WA) and AS-OCT (Fourier domain OCT CASIA2, Tomey Technology and vision, Germany).

Central corneal endothelial photographs are taken with the Topcon SP-IP specular microscope (Topcon Europe B.V., Capelle a/d Ijssel, the Netherlands) and total ocular wavefront is measured with iTrace (Tracey Technologies, Inc.).

Ocular discomfort is subjectively evaluated in each eye by a specific visual analogous rating scale at 4h, 8h, 12h, 24h and thereafter daily up to 1 week postoperatively.

All the above mentioned examinations are repeated at 1, 3, 6, 12 and 24 months after treatment. At 1 day and 1 week after treatment, solely UCVA, Auto refractor measurements, slit-lamp examination are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for corneal crosslinking.
* Progressive keratoconus documented with a consistent decrease of best corrected visual acuity with no other explanation, an unquestionable historical progression, or a progression documented with the Pentacam Scheimpflug camera with at least 2 of the following: progressive anterior and/or posterior corneal steepening and/or progressive corneal thinning and/or increased rate of corneal thickness change from the periphery to the center.
* A keratoconus diagnosis based on abnormal posterior elevation, abnormal corneal thickness distribution and clinical noninflammatory corneal thinning using the "Belin/Ambrósio enhanced ectasia" measurements of the Pentacam Scheimpflug camera.
* Minimum corneal thickness of 400 µm at the thinnest point before epithelial removal.
* 18-35 years of age
* No ocular abnormalities except keratoconus
* No previous ocular surgery
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* Age under 18 or over 35
* Any corneal abnormalities except keratoconus
* Pregnancy or lactation
* Previous ocular surgery
* Cognitive insufficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | 1, 3, 6, 12 and 24 months after treatment.
  Change from baseline in Uncorrected Distance Visual Acuity
Keratometry readings | 1, 3, 6, 12 and 24 months after treatment
  Change from baseline in Keratometry readings, Kmean (average), K1 (flat meridian), K2 (steep meridian) and Kmax (steepest radius of curvature) assessed with the Pentacam HR Scheimpflug camera

SECONDARY OUTCOMES:
Subjective Ocular Discomfort Scores | 4, 8h and 1, 2, 3, 4, 5, 6 and 7 days after treatment.
  Change in a Ocular Discomfort Visual Analogous Scale after treatment.
Manifest Refractive Spherical Equivalent (MRSE) | 1, 3, 6, 12 and 24 months after treatment.
  Change from baseline in Manifest Refractive Spherical Equivalent
Corneal Endothelial cell density (ECC) | 12 and 24 months after treatment
  Change from baseline in corneal endothelial cell density
Best Spectacle Distance Visual Acutiy (BSCVA) | 1, 3, 6, 12 and 24 months after treatment.
  Change from baseline in Best Spectacle Distance Visual Acutiy

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, Principal Investigator — Department of Clinical Sciences/Ophthalmology, Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No